CLINICAL TRIAL: NCT04454242
Title: Comparison of the Effects of High and Low Intensity Expiratory Muscle Strength Training in Patients With Obstructive Sleep Apnea Syndrome
Brief Title: High and Low Intensity Expiratory Muscle Strength Training in Patients With Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evren Chest and Cardiovascular Surgery Education and Research Hospital (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, NUREL ERTURK, Clinical Physiotherapist, Ahi Evren Chest and Cardiovascular Surgery Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020/09
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-01

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Expiratory muscle strength training; Snoring; Sleep quality; EMST
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-EMST (Experimental): At 30% of the maximum expiratory pressure (MEP), 25 breaths, 7 days / week, a total of 8 weeks will be trained once a day with a 1-minute rest cycle in 5 breaths.
  Patients will be invited to control every 2 weeks. MEP measurements will be repeated and the training value will be adjusted in 30% of the new measurement.
  Interventions: Other: Expiratory muscle trainig
- H-EMST (Active Comparator): In 60% of the maximum expiratory pressure (MEP), 25 breaths a day, 7 days / week, a total of 8 weeks will be trained with a 1-minute rest cycle in 5 breaths.
  Patients will be invited to control every 2 weeks. MEP measurements will be repeated and the training value will be adjusted in 60% of the new measurement.
  Interventions: Other: Expiratory muscle trainig

INTERVENTIONS:
Other: Expiratory muscle trainig — This exercise will be used to strengthen forced expiratory muscles.

SUMMARY:
The effect of expiratory muscle strength training (EMST) on sleep quality, disease severity, and respiratory muscle strength has been previously investigated in OSA syndrom. Only the effects of the high-intensity short-term EMST study in moderate OSAS patients were studied. High intensity and low intensity EMST has advantages and disadvantages.The study aims to compare the effects of high (60% MEP) and low (30% MEP) expiratory muscle strength training (EMST) on disease severity, sleep efficiency, snoring, fatigue severity and quality of life in severe OSAS patients.

DETAILED DESCRIPTION:
Ahi Evren Chest Cardiovascular Surgery Training Research Hospital In sleep lab, polysomnography will be directed to the physiotherapist by the pulmonologist with severe OSAS patients. Patients will be divided into two groups by block randomization method. The study was planned as double-blind. Patients will not know what treatment they are receiving, the doctor does not know what treatment the patient is receiving, and technicians who take and analyze polysomnography will not know what treatment the patients are receiving.

Severe OSAS patients with MEP 30% (low intensity) to the first group, MEP 60% (high intensity) to the second group with expiratory muscle training device, 7 days / week, 25 breaths per day, 1 minute rest for 5 breaths will be run with the cycle. The training will take a total of 8 weeks. The follow-up of the patients will be done remotely by phone. MEP measurements will be repeated every 2 weeks in the hospital and the new training workload will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with severe OSAS by Polysomnography in Ahi Evren Chest, Cardiovascular Surgery Training and Research Hospital Sleep Center will be included.
2. General health condition is stable

Exclusion Criteria:

1. Passed stroke,
2. Neurological disease and psychological disease
3. Cardiac disease
4. Hypothyroidism
5. Serious obstructive nasal disease,
6. A history of infection in the past month.
7. Previous oroferengeal surgery history
8. With a BMI of 40 kg / m2 or more,
9. Using substance, alcohol, sedative and hypnotic drugs

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Disease severity | 2 day
  Polysomnography recordings will be taken especially sleep efficiency and apnea-hypopnea index (AHI). Higher sleep efficiency and lower AHI values shows that patient have better status and lower disease severity
Respiratory muscle strength | 5 day
  Maximal inspiratory and expiratory muscle strength measurement with mouth pressure device

SECONDARY OUTCOMES:
Daytime sleepiness | 2 day
  Epworth Sleepiness Scale (ESS). Minimum and maximum scores: 0-24. The higher ESS score means the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'
Snoring severitiy and frequency | 2 day
  Berlin Questionnaire: Snoring frequency (0-3) and severity (0-4). Higher scores show higher snoring frequency and severity.
Sleep quality | 2 day
  The Pittsburgh Sleep Quality Index (PSQI). Minimum and maximum scores: 0-21. Higher PSQI scores show worse sleep quality.
Fatigue severity. | 2 day
  Fatigue Severity Scale (FSS) . Minimum and maximum scores: 0-7. FSS scores higher than 4 shows high intensity fatigue perception

OTHER OUTCOMES:
Antropometric measurements | 2 day
  Neck circumference, Waist circumference, Hip circumference, Waist to hip ratio with circumference measurement method

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik-Kutukcu, PhD, Study Director — Hacettepe University
Locations (1):
- Trabzon Ahi Evren Thoracic and Cardiovascular Surgery Training and Research Hospital, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No